CLINICAL TRIAL: NCT04770766
Title: Implementation of the Non-medical Practitioner Workforce Into the Urgent and Emergency Care System Skill-mix in England: a Mixed Methods Study of Configurations and Impact
Brief Title: Non-medical Practitioner Workforce in the Urgent and Emergency Care System Skill-mix in England
Acronym: SKILLmix-ED
Status: Completed | Type: Observational
Sponsor: Kingston University (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government); St George's University Hospitals NHS Foundation Trust (Other); Surrey and Sussex Healthcare NHS Trust (Other); University of Surrey (Other); Royal Holloway University (Other)
Responsible Party: Sponsor
Other Study IDs: NIHR131356
Record Dates: First submitted 2021-02-12; First posted 2021-02-25 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Emergencies
Keywords: Emergency Service, Hospital; Workforce; Professional Autonomy; non-medical practitioners; Health Services Research
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (7):
- Staff observation: Doctor-in-training and non-medical practitioner volunteers
  Interventions: Other: Non-medical practitioners
- Patient questionnaires: Patients attending the Emergency Department of one of six NHS trusts participating in the research as a case study
  Interventions: Other: Non-medical practitioners
- Case study NHS Trusts: NHS organisations with an Emergency Department participating as a case study site
  Interventions: Other: Non-medical practitioners
- All England NHS Trusts: NHS Trusts whose Emergency Department (n=183) records data is held by NHS Digital and will be provided anonymously/without individual patient consent (these anticipated hundreds of thousands of records are not included in the enrolled patient numbers)
  Interventions: Other: Non-medical practitioners
- Patient interviews: Patients attending the Emergency Department of one of six NHS trusts participating in the research as a case study and volunteering to take part in an interview following completion of the patient questionnaire
  Interventions: Other: Non-medical practitioners
- Staff interviews: Staff working in the Emergency Department of one of six NHS trusts participating in the research as a case study and volunteering to take part in an interview
  Interventions: Other: Non-medical practitioners
- Stakeholder interviews: Senior NHS clinicians, managers, commissioners and lay representatives with roles and interests in the non-medical practitioner workforce
  Interventions: Other: Non-medical practitioners

INTERVENTIONS:
Other: Non-medical practitioners — All observational research activity in each cohort is related to the exposure of non-medical practitioners in the Emergency Department or Urgent Treatment Centre

SUMMARY:
This study will explore the result of different skill-mix in ED/UTCs in England, to make recommendations about the best balance.

Patient and public involvement (PPI) representatives have helped design the study. There will be an independent PPI panel who can feed in their views and experiences to all parts of the study. The panel will be run by an experienced patient and public involvement expert, who is a member of the core study team.

The study will be split into four phases over two-and-a-half years.

Phase One will find out in detail what the staffing models are in EDs/UTCs. The investigators will look at published research evidence and at NHS public documents, and will interview regional and national senior NHS clinicians, managers, commissioners and lay representatives. Then, information about staff which is already collected regularly across England will be analysed for patterns. What non-medical practitioners do and how independently they work in two different ED/UTCs will also be examined. The panel of patient and public involvement representatives and a panel of non-medical practitioners will help interpret these findings. The study will develop a system for classifying 'skill-mix' in each organisation and a way to measure how much support and supervision non-medical practitioners need.

Phase Two will look at figures regularly collected from all NHS Trusts in England between 2017 and 2021, to assess whether different skill mixes lead to different patient outcomes. The number of patients who return again to the ED within a week is the primary outcome.

Phase Three will involve looking in detail in six ED/UTCs. The investigators will collect in depth local data to add to the national data we looked at in Phase Two. This will include looking closely at staff records and patients' clinical records to illustrate more detail about skill-mix in the organisations and the outcomes for patients. The study plans to gauge how independently the types of practitioners assess and treat patients and to also survey and interview patients so that their experience can be understood, alongside the views of staff who will also be interviewed.

Phase Four will pull all of the results together. The panels of patient and public involvement representatives and non-medical practitioners will help with this synthesis. The study aims to make recommendations on skill-mix and levels of independence that will deliver the best outcomes for patients, for staff and for the NHS.

DETAILED DESCRIPTION:
Primary research question

What is the impact of different non-medical practitioner skill-mix in Emergency Departments (ED) and Urgent Treatment Centres (UTC) in acute hospitals on patient and service processes and outcomes?

Background

Increasing demand for emergency and urgent care has occurred alongside staffing shortage, particularly of doctors. Re-shaping of the workforce has resulted, including the introduction of non-medical practitioners (NMPs), such as nurse practitioners and physician associates. Despite 20 years of NMPs in EDs, there is limited evidence of effectiveness of individual roles, and none as to appropriate skill-mix of staff, at what level of independence from senior medical staff.

Aim

To explore how NMPs are being deployed and the impact of different skill-mix including NMPs in EDs and UTCs on patient experience, quality of care, clinical outcomes, activity, staff experience and costs in acute NHS trusts in England, in order to inform workforce decisions of clinicians, managers and commissioners.

Methods

A mixed methods study will be conducted in three phases.

Phase One (months 1-12) aims to describe the rationale for, and configurations of, the NMP workforce in EDs/UTCs in England, and to develop analytical tools.

* The investigators will undertake and publish a scoping literature and policy review on NMP development and skill-mix outcomes, informed by interviews with senior NHS clinicians, managers, commissioners and lay representatives (Work package [WP] 1)
* NHS Digital and NHS Benchmarking national data, 2017-2021 will be used to describe quantitatively the NMP and other clinical workforce (skill-mix); and observation (WP2) will enable qualitative description of the level of independence/supervision of NMPs and doctors.
* WP1 and WP2 results will be triangulated in consultative activities with patient and public and NMP representatives, and the independent study steering committee, to develop three analytical tools: a skill-mix ratio classification, a quantitative measure of independence and supervision, and a logic model for NMP skill-mix (WP3).

Phase two (months 13-18) aims to utilise the analytical tools to assess the impact of skill-mix ratios on national ED/UTC indicators of quality.

•The investigators will conduct and publish a quasi-experimental study of associations of skill-mix ratio classifications with our primary outcome (rate of unplanned return to the ED/UTC in seven days, a proxy for clinical safety), secondary outcomes (national indicators of ED/UTC quality and performance), and cost-effectiveness. (WP4)

Phase three (months 13-24) aims to explain the effectiveness and acceptability of skill-mix ratios through investigation in six local-level case study sites.

* The WP4 analysis will be repeated with added precise local quantitative data on NMP types (trust management information), controlling for level of independence/supervision of the clinician (collected via structured observation). Patient satisfaction will be added as an outcome, collected prospectively via questionnaire (WP5).
* The experience of including NMPs in the skill-mix will be investigated through qualitative interviews with patients and staff (WP6).

In Phase four (months 25-30) the investigators will prepare a synthesis of findings, using the logic model, for structured discussion at a stakeholder event to prepare recommendations and outputs.

Timelines for delivery

The study will take place from March 2021 to August 2023.

Anticipated impact and dissemination

The research will generate new knowledge and understanding of optimum/most effective/impact of different skill-mix outcomes to translate into workforce models with our NHS partners. Commissioners, clinicians and managers will be able to assess their local skill-mix in relation to the guidance on (optimum) skill-mix outcomes. Dissemination throughout the study will include policy briefings, academic outputs, bite-size findings, conference presentations and social and mainstream media routes accessible to stakeholders.

ELIGIBILITY:
Inclusion Criteria:

* All NHS trusts: - all in England
* Case study trusts: six NHS trusts in England exhibiting different non-medical practitioner to other clinician skill-mix ratios, and giving board-level consent to participation
* Stakeholders: senior NHS clinicians, managers, commissioners and lay representatives with roles and interests in the non-medical practitioner workforce
* Staff observation: non-medical practitioners and junior doctors-in-training in one of six NHS case study trusts who volunteer to being observed in practice for specified time periods
* Staff interviews: staff working with non-medical practitioners and junior doctors-in-training in one of six NHS case study trusts who volunteer to be interviewed
* Patient questionnaire: patients attending the Emergency Department in one of the six NHS case study trusts during specified study data collection periods who agree to take a questionnaire for completion
* Patient interviews: patients attending the Emergency Department in one of the six NHS case study trusts during specified study data collection periods who return a completed questionnaire and volunteer to be interviewed

Exclusion Criteria:

* Patient data outside of the study time periods
* Staff or patient volunteers in sub-groups (e.g. personal characteristics or roles) that are already represented /over-represented amongst volunteer participants
* those for whom English is difficult to understand or speak/do not have someone with them who can interpret or support.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study population varies for each of the study components, but is encompassed within the following:
  * patients attended at Emergency Departments and Urgent Treatment Centres in England 2017-2022
  * staff working closely with and stakeholders to the non-medical practitioner workforce in Emergency Departments and Urgent Treatment Centres in England
Sampling Method: Non-Probability Sample
Enrollment: 840 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Re-attendance | 7 days
  Re-attendance at the Emergency department following the index event

SECONDARY OUTCOMES:
Left without being seen | up to 8 hours
  Left Emergency Department before being seen for treatment
Time to initial assessment | Up to 8 hours
  Time from patient arrival to being assessed by a clinician
Time to treatment | Up to 8 hours
  Time from patient arrival to being treated by a clinician
Total time | Up to 8 hours
  Time from patient arrival to leaving the Emergency Department
Clinical investigation | Up to 8 hours
  Clinical investigations recorded by the attending clinician in the Emergency Department
Treatment code | Up to 8 hours
  Treatments recorded using a code by the attending clinician in the Emergency Department
Onward referral /treatment complete | Up to 8 hours
  Patient's next destination recorded in the Emergency Department
Cost | 1 hour
  Staff unit costs

OTHER OUTCOMES:
Stakeholder perspectives | Up to 6 months
  Qualitative exploration of the factors and rationale influencing current and future ED/UTC workforce configurations and the inclusion of different types of NMPs
Staff perspectives | 3 months
  Qualitative exploration of views of staff closely related to working with NMPs
Patient satisfaction | 1 and 28 days
  Quantitative measure of patient experience of being attended in Emergency Departments with differing skill-mix ratios
Patient perspectives | 28 days
  Qualitative exploration of views of patients attended in Emergency Departments with differing skill-mix ratios

CONTACTS AND LOCATIONS:
Overall Officials: Mary Halter, PhD, Principal Investigator — Kingston University
Locations (2):
- United Kingdom (2):
  - St George's University Hospital NHS Foundation Trust, London, London
  - Faculty of Health, Science, Social Care and Education, Kingston, Surrey

IPD SHARING:
Plan to Share IPD: No